CLINICAL TRIAL: NCT00130208
Title: The Collaborative Study Group Trial: The Effect of Sulodexide in Patients With Type 2 Diabetes and Microalbuminuria
Brief Title: Effect of Sulodexide in Early Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Collaborators: Collaborative Study Group (CSG) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KRX-101-301
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetes; Diabetes Mellitus, Type 2; Albuminuria; Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Diabetes Mellitus, Type 2; Albuminuria | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulodexide (Experimental): Also known as KRX-101. All patients will be on standard of care ACE or ARBs.
  Interventions: Drug: Sulodexide
- Placebo (Placebo Comparator): All patients will be on standard of care ACE or ARBs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulodexide — 100 mg sulodexide gelcaps
  Other Names: KRX-101
  Arms: Sulodexide
Drug: Placebo — 0 mg gelcap
  Other Names: Placebo oral gelcap
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether treatment with sulodexide is effective in reducing the level of urine albumin excretion in patients with early diabetic kidney disease expressed as microalbuminuria.

DETAILED DESCRIPTION:
Diabetic nephropathy is an important cause of morbidity and mortality in patients with either type 1 or type 2 diabetes mellitus. The pathogenesis and natural history of diabetic nephropathy is characterized initially by microalbuminuria followed by a progressive decline in glomerular function. An emerging body of evidence supports the notion that glomerular capillary wall and mesangial alterations in diabetic nephropathy involve pathobiochemical alterations of glycoproteins in these structures. Evidence, in experimental animals rendered diabetic, reveals that the administration of heparin and other anionic glycoproteins (GAG) can effectively prevent the biochemical alterations which are responsible for albuminuria. Sulodexide, an orally active agent which does not have anticoagulant properties associated with its oral dose range, is comprised of three naturally occurring glycosaminoglycan (GAG) polysaccharide components isolated from porcine intestinal mucosa. Small clinical studies employing sulodexide, have shown that albuminuria is significantly diminished in patients with diabetic nephropathy, even when these patients are receiving angiotensin II receptor blockers (ARB) or angiotensin converting enzyme inhibitors (ACEI), agents already proven to reduce albuminuria and slow progressive diabetic nephropathy.

This study is designed to evaluate whether sulodexide is safe and effective in treating subjects with type 2 diabetic nephropathy. Subjects with type 2 diabetes and microalbuminuria (defined as a urinary albumin to creatinine ratio,(ACR)in men 35-200 mg/G and in women 45-200 mg/G) who are also receiving either irbesartan 300 mg/day, losartan 100 mg/day, or a maximum approved dose of an angiotensin receptor blocker (ARB) or angiotensin converting enzyme inhibitor (ACEI) will be enrolled in the study. The study will consist of the following periods:

* Screening: of 1-2 weeks for assessing basic eligibility/exclusion criteria
* Run-in: of up to 16 weeks on maximal dose of ARB or ACE with stable blood pressure control
* Qualifying visit: qualifying patients are on maximal dose of ARB or ACE for a minimum of 4 months with stable BP control, SBP <150 mmHg, DBP <90 mmHg and albumin to creatinine ratio, (ACR) between in men 35-200 mg/G and in women 45-200 average of 3 first morning voids
* Randomization: patients are randomized to sulodexide 100 mg or matching placebo administered orally twice a day.
* Maintenance: 26 week maintenance period, with 4 visits to monitor safety and ACR
* Washout Period: 8 week washout period, with 2 visits to monitor safety and ACR

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Serum creatinine equal to or less than 1.5 mg/dL
* Microalbuminuria, defined by a urine albumin/creatinine ratio in men; 35- 200 mg albumin/G creatinine, in women; 45-200 mg albumin/G creatinine
* Blood pressure controlled to less than 150/90 mmHg
* Willing to change antihypertensive medication regimen if necessary

Exclusion Criteria:

* Age of onset of type 2 diabetes <18 years;
* HbA1C >10.0%;
* Morbid obesity defined as a body mass index (BMI) >= 45 kg/m2;
* Type 1 (insulin-dependent; juvenile onset) diabetes;
* Renal disease as follows:

  * Patients with known non-diabetic renal disease
  * Renal allograft
* Absolute requirement for combination therapy of angiotensin converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARB);
* Cardiovascular disease as follows:

  * Unstable angina pectoris within 3 months of study entry;
  * Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty or stent placement within 3 months of study entry;
  * Transient ischemic attack within 3 months of study entry;
  * Cerebrovascular accident within 3 months of study entry;
  * Symptomatic heart failure requiring ACE inhibition;
  * New York Heart Association Functional Class III or IV heart failure;
  * Obstructive valvular heart disease or hypertrophic cardiomyopathy;
  * Second or third degree atrioventricular block not successfully treated with a pacemaker
* Need for chronic (>2 weeks) immunosuppressive therapy, including corticosteroids (excluding inhaled or nasal steroids);
* History of multiple drug allergies;
* New diagnosis of cancer or recurrent cancer within 5 years of screening ( (except non-melanoma skin cancer);
* Psychiatric disorder that interferes with the patient's ability to comply with the protocol;
* Inability to tolerate oral medication or a history of significant malabsorption;
* Inability to remain on a stable dose of the following class of medications 30 days prior to randomization and throughout the study:

  * 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors (statins);
  * Peroxisome proliferator-activated receptor gamma (PPAR gamma inhibitors (glitazones);
  * Cyclooxygenase-2 inhibitors (COX-2 inhibitors); or
  * Non-steroidal anti-inflammatory drugs (NSAIDS);
* History of alcohol or other drug abuse within 12 months of study entry;
* Known human immunodeficiency virus (HIV) disease;
* Any other medical condition which renders the patient unable to or unlikely to complete the study, or which would interfere with optimal participation in the study or produce significant risk to the patient;
* Receipt of any investigational drugs (including placebo) within 30 days of enrollment;
* Evidence of hepatic dysfunction including total bilirubin >2.0 mg/dL or liver transaminase (AST or ALT) >3 times upper limit of normal;
* Anticipated surgery within trial period;
* Inability to cooperate with study personnel or history of noncompliance to medical regimen (i.e., patients who would be expected to comply poorly with treatment);
* Known allergies or intolerance to any heparin-like compound;
* Untreated urinary tract infection that would impact urinary protein values; or
* Prior exposure to sulodexide, either in a clinical setting or as a participant in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2005-08; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund J Lewis, M.D., Study Director — The Collaborative Study Group, Rush University Medical Center, Chicago, IL USA; Robert C Atkins, M.D., Principal Investigator — The Collaborative Study Group, Monash Medical Center, Clayton, Victoria, AUSTRALIA; Dick deZeeuw, M.D., Principal Investigator — The Collaborative Study Group, University of Groningen, NETHERLANDS; Itamar Raz, M.D., Principal Investigator — The Collaborative Study Group, Hadassah University, Jerusalem, ISRAEL
Locations (3):
- The Collaborative Study Group, Clinical Coordinating Center for U.S. and Canadian Clinics, Rush University Medical Center, Chicago, Illinois, United States
- The Collaborative Study Group, Clinical Coordinating Center for the Pacific Region, Monash Medical Center, Melbourne, Victoria, Australia
- The Collaborative Study Group, Clinical Coordinating Center for European Clinics, University of Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis EJ, Lewis JB, Greene T, Hunsicker LG, Berl T, Pohl MA, de Zeeuw D, Heerspink HL, Rohde RD, Atkins RC, Reutens AT, Packham DK, Raz I; Collaborative Study Group. Sulodexide for kidney protection in type 2 diabetes patients with microalbuminuria: a randomized controlled trial. Am J Kidney Dis. 2011 Nov;58(5):729-36. doi: 10.1053/j.ajkd.2011.06.020. Epub 2011 Aug 26. PMID 21872376

RESULTS

PARTICIPANT FLOW:
Period: Maintenance Period (26 Weeks)
Arm/Group | Sulodexide | Placebo
Started | 524 | 532
Valid Albumin Creatinine Ratio (Valid albumin creatinine ratio at baseline and week 26) | 492 | 494
Completed | 500 | 502
Not Completed | 24 | 30
Not completed — Adverse Event | 10 | 12
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Lost to Follow-up | 5 | 4
Not completed — Other | 1 | 1
Period: Washout Period (8 Weeks)
Arm/Group | Sulodexide | Placebo
Started | 500 | 502
Completed | 494 | 490
Not Completed | 6 | 12
Not completed — Adverse Event | 3 | 6
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulodexide | Placebo | Total
Number analyzed (Participants) | 524 | 532 | 1056
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (9.73) | 62.3 (9.90) | 62.2 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 124 | 254
  Male | 394 | 408 | 802
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 31 | 59
  Not Hispanic or Latino | 496 | 501 | 997
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 33 | 34 | 67
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 39 | 28 | 67
  White | 440 | 451 | 891
  More than one race | 8 | 15 | 23
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Conversion From Microalbuminuria to Normoalbuminuria
Description: The primary efficacy variable was the fraction of those patients in the ITT population with valid baseline and Week 26 ACRs in whom "therapeutic success" was achieved at Week 26 measured as a conversion of microalbuminuria to normoalbuminuria and at least a 25% reduction in ACR relative to baseline
Time Frame: 26 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sulodexide | Placebo
Number analyzed (Participants) | 492 | 494
Participants | 39 | 30

2. Primary Outcome: Number of Subjects With Greater Than 50% Reduction in Microalbuminuria
Description: During the treatment period, KRX-101 is being compared to placebo to assess whether a 50% reduction in microalbuminuria has been achieved.
Time Frame: 26 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sulodexide | Placebo
Number analyzed (Participants) | 492 | 494
Participants | 76 | 87

3. Secondary Outcome: Change in Serum Albumin From Baseline to End of 26 Weeks
Time Frame: 26 Weeks
Population: Participant numbers include those with both baseline and week 26 measurements
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Sulodexide | Placebo
Number analyzed (Participants) | 489 | 496
percent change | -0.02 (0.01) | -0.02 (0.01)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the full duration of the trial (34 weeks)
Description: The safety population consisted of all patients who were administered at least 1 dose of study medication. There was one patient in the sulodexide group who was randomized but did not receive study medication
Arm/Group | Sulodexide | Placebo
All-Cause Mortality (participants affected / at risk) | 2/523 | 3/532
Serious Adverse Events (participants affected / at risk) | 21/523 | 33/532
Other Adverse Events (participants affected / at risk) | 348/523 | 358/532
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sulodexide (N=523) | Placebo (N=532)
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Post-procedural hematoma (Blood and lymphatic system disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 1
Aortic Stenosis (Cardiac disorders) | 1 | 0
Aortic Aneurysm (Cardiac disorders) | 1 | 0
Transient ischemic attack (Cardiac disorders) | 1 | 0
Diabetic Foot (Metabolism and nutrition disorders) | 1 | 0
Pancreatitis (Infections and infestations) | 1 | 0
Device Failure (Injury, poisoning and procedural complications) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Death (General disorders) | 0 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 3
Coronary artery disease (Cardiac disorders) | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sigmoiditis (Infections and infestations) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal Cord Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid Artery Stenosis (Cardiac disorders) | 0 | 1
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkins Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Hemorhage Intracranial (Nervous system disorders) | 0 | 1
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulodexide (N=523) | Placebo (N=532)
Coronary Artery Disease (Cardiac disorders) | 6 | 3
Diarrhea (Gastrointestinal disorders) | 21 | 20
Constipation (Gastrointestinal disorders) | 10 | 11
Nausea (Gastrointestinal disorders) | 10 | 6
Abdominal Pain (Gastrointestinal disorders) | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 6
Edema Peripheral (General disorders) | 55 | 65
Edema (General disorders) | 13 | 12
Chest Pain (General disorders) | 8 | 6
Asthenia (General disorders) | 9 | 4
Fatigue (General disorders) | 4 | 9
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 18 | 24
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 21 | 18
Urinary Tract Infection (Infections and infestations) | 16 | 20
Bronchitis (Infections and infestations) | 9 | 16
Influenza (Infections and infestations) | 8 | 12
Sinusitis (Infections and infestations) | 9 | 5
Gastroenteritis (Infections and infestations) | 3 | 6
Cardiac Murmur (Investigations) | 5 | 9
Weight Increased (Investigations) | 6 | 4
Blood glucose increased (Investigations) | 1 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 17
Pain in extremities (Musculoskeletal and connective tissue disorders) | 11 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 13
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 9
Headache (Nervous system disorders) | 16 | 17
Dizziness (Nervous system disorders) | 13 | 15
Hypoesthesia (Nervous system disorders) | 2 | 6
Depression (Psychiatric disorders) | 2 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Rales (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 9
Hypertension (Vascular disorders) | 12 | 15
Hypotension (Vascular disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No